CLINICAL TRIAL: NCT06791980
Title: Association Between Pro-inflammatory Cytokines and Depressive Symptoms in Patients with Rheumatoid Arthritis: Evaluating the Impact of an Integrated Care Approach
Brief Title: Integrated Care Approach for Rheumatoid Arthritis Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Tzung-Yi Tsai, Researcher, Dalin Tzu Chi General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B11204006
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Routine care (Other): This consisted of consultation about disease symptoms, related treatments, and conventional disease management.
  Interventions: Other: CM-TCM

INTERVENTIONS:
Other: CM-TCM — To assess the long-term effects of integrated case management model involving traditional Chinese medicine (CM-TCM) model. The persons participating will be invited to enroll in this stage, and they will be assigned to receive either the usual care or a usual care plus integrated 3-month CM-TCM

SUMMARY:
The goal of this study is to learn about the long-term effects of integrated care approach in persons over the age of 20 who take part in integrated care approach to treat their rheumatoid arthritis (RA). The main question is to explore whether adding the integrated care approach into routine care can lower pro-inflammatory cytokines and depressive symptom in RA persons over age 20 when taken long-term to treat RA?

ELIGIBILITY:
Inclusion Criteria:

age of at least 20 years; willingness to participate in the survey; having the physician-diagnosed RA with the International Classification of Diseases, 9th Revision, Clinical Modification code of 714.0

Exclusion Criteria:

* having physician-based diagnosis of cognitive impairment and with the ability to express opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
cytokines | From enrollment to the end of treatment at 12 weeks"
  Serum cytokine levels contained interleukin (IL)-6, IL-1, IL-17 and tumor necrosis factor (TNF)-alpha,

SECONDARY OUTCOMES:
depressive symptom | From enrollment to the end of treatment at 12 weeks"
  It is measured by self-reported scale

CONTACTS AND LOCATIONS:
Locations (1):
- Dalin Tzuchi Hospital, Chiayi City, Chiayi, Taiwan

IPD SHARING:
Plan to Share IPD: No